CLINICAL TRIAL: NCT02402933
Title: A Multiple Center, Open Label, Prospective Study to Evaluate the Effectiveness and Ease-Of-Use of AMG504-1 Administered in the Home or School Environments for Treating Hypoglycemia in Children and Adolescents With T1D
Brief Title: Clinical Usability of Nasal Glucagon in Treatment of Hypoglycemia in Children and Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16423; I8R-MC-B001 (Other: Eli Lilly and Company); AMG109 (Other: Locemia Solutions ULC)
Record Dates: First submitted 2015-03-25; First posted 2015-03-30 (Estimated); Results first posted 2017-06-26 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Hypoglycemia; Diabetes Mellitus
MeSH Terms: conditions — Hypoglycemia; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nasal Glucagon (Experimental): A single dose of 3mg glucagon nasal powder administered using a nasal powder delivery device for the treatment of moderate or severe hypoglycemic events; a maximum of 4 events per participant during the study.
  Interventions: Drug: Nasal Glucagon

INTERVENTIONS:
Drug: Nasal Glucagon — 3 mg nasal glucagon powder
  Other Names: Dry-Mist nasal glucagon; AMG504-1; LY900018

SUMMARY:
Up to fifty (50) children and adolescents with type 1 diabetes (T1D) aged 4 to ˂18 years at time of enrolment will be selected for inclusion in the study. The target is to obtain treatment response and user-experience data following use of Nasal Glucagon (LY900018) in treating episodes of hypoglycemia.

DETAILED DESCRIPTION:
This study is designed to evaluate the effectiveness of nasal glucagon (NG) administered under clinical use conditions in treating episodes of moderate or severe hypoglycemia in persons with T1D.

This study also aims to assess the ease with which caregivers can administer the experimental medication in treatment of hypoglycemic events.

ELIGIBILITY:
Inclusion Criteria:

* Availability for the entire study period.
* Motivated Child/Adolescent with diabetes (C/AWD) and caregiver(s) and absence of intellectual problems likely to limit the validity of consent to participate in the study or the compliance with protocol requirements; ability to cooperate adequately; ability to understand and observe the instructions of the qualified investigator or designee.
* C/AWD lives with one or more caregivers who are available to administer the glucagon in case of an episode of severe or moderate hypoglycemia.
* Male or female C/AWD with a history of type 1 diabetes >1 year.
* C/AWD aged of at least 4 years of age but less than 18 years.
* A female C/AWD must meet one of the following criteria:

  a) Participant is of child-bearing potential and agrees to use one of the accepted contraceptive regimens throughout the entire duration of the study (from the pre-trial evaluation and enrollment visit until study completion). An acceptable method of contraception includes one of the following: (i) Abstinence from heterosexual intercourse (ii) Systemic contraceptives (birth control pills, injectable/implantable/ insertable hormonal birth control products, transdermal patch) (iii) Intrauterine device (iv) Condom with spermicide, OR b) Participant is of non-child-bearing potential, defined as a female who had had a hysterectomy or tubal ligation, is clinically considered infertile or has not yet reached menarche.
* In good general health with no conditions that could influence the outcome of the trial, and in the judgment of the Investigator is a suitable candidate for the study based on review of available medical history, physical examination and clinical laboratory evaluations.
* Willingness to adhere to the protocol requirements.

Exclusion Criteria:

* Females who are pregnant according to a positive urine pregnancy test, actively attempting to get pregnant, or lactating.
* History of significant hypersensitivity to glucagon, or any related products as well as severe hypersensitivity reactions (such as angioedema) to any drugs.
* Presence of cardiovascular, gastrointestinal, liver or kidney disease, or any other conditions which in the judgment of the investigator could interfere with the absorption, distribution, metabolism or excretion of drugs or could potentiate or predispose to undesired effects.
* Presence or history of pheochromocytoma (i.e. adrenal gland tumor) or insulinoma.
* Use of daily systemic beta-blockers, indomethacin, warfarin or anticholinergic drugs.
* Concomitant maintenance therapy with any drug that would influence the outcome of the trial, at the discretion of the Investigator and the Sponsor.
* Regular consumption of 3 or more units of alcoholic beverages per day.
* Current participation in another clinical trial, intent to enroll in another clinical trial during this clinical study or use of an Investigational Product (in another clinical trial) within the prior 30 days.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2015-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - Private Clinic, Tallahassee, Florida
  - Private Clinic, Baltimore, Maryland
  - New England Diabetes and Endocrinology Center (NEDEC), Waltham, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants and their principal caregiver(s) (such as parents, family member, roommate, teacher, and coach) were trained in the use of nasal glucagon.
Groups:
- Nasal Glucagon (NG): A single dose of 3 mg glucagon nasal powder administered using a nasal powder delivery device for the treatment of moderate or severe hypoglycemic events; a maximum of 4 events per participant during the study.
Period: Overall Study
Arm/Group | Nasal Glucagon (NG)
Started | 26
Received at Least One Dose of Study Drug | 22
Completed | 12
Not Completed | 14
Not completed — Withdrawal by Subject | 4
Not completed — Discontinued; Site Termination | 10

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Nasal Glucagon (NG): Nasal glucagon 3 milligram (mg)
Arm/Group | Nasal Glucagon (NG)
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.7 (3.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Awakening or Returning to a Normal Status Within 30 Minutes Following Studied Drug of Administration
Description: Responses to questions completed by the caregiver are used to assess this outcome. An episode of severe hypoglycemia is generally defined as an event associated with severe neuroglycopenia usually resulting in coma or seizure and requiring parenteral therapy (glucagon or intravenous glucose) administered by a third party. In this study moderate hypoglycemia is defined as an episode wherein the child/adolescent with diabetes has symptoms and/or signs of neuroglycopenia and has a blood glucose ≤3.9 millimoles per liter (mmol/L) (70 milligram per deciliter [mg/dL]) based on a blood sample taken at or close to the time of treatment.
Time Frame: Within 30 minutes after each drug administration for an episode of hypoglycemia
Population: Participants who received at least 1 dose of NG with evaluable treatment response. Events for which participants required external professional medical assistance or used injected glucagon or oral carbohydrates within 30 minutes and before responding were non-evaluable. The good clinical practice (GCP) non-compliant site were also excluded.
Measure: Number; unit: participants
Groups:
- Nasal Glucagon: Nasal glucagon (NG) 3 mg
Arm/Group | Nasal Glucagon
Number analyzed (Participants) | 14
participants | 14

2. Secondary Outcome: Assessment of Ease-of-use of Dry-Mist Nasal Glucagon by Completion of Questionnaire by the Caregiver
Description: Assess ease-of-use of intranasal administered glucagon in the hands of caregivers of participants who may be called upon to treat episodes of hypoglycemia.
  Measurement for Degree of difficulty: opening the kit, Degree of difficulty: understanding the instructions on how to use the kit, Degree of difficulty: administering the medication into the nostril, Degree of satisfaction is 1 (Very Difficult) to 7 (Very Easy). Measurement for Dry Mist Nasal Glucagon will be easy to teach other caregivers, Nasal formulation of glucagon is less intimidating for caregivers, Dry Mist Nasal Glucagon is easy to carry and would be willing to carry it, Intranasal delivery of glucagon is preferable: level of agreement 1 (Strongly Disagree) to 7 (Strongly Agree).
Time Frame: After each drug administration for an episode of hypoglycemia
Population: Participants who received at least 1 dose of NG and experienced at least 1 hypoglycemic event. Participants from the GCP non-compliant site were excluded. Proportions and n are based on the total number of hypoglycemic events (N=33) of 14 participants; except "Compare to Injectable" is based on 8 events.
Measure: Count of Units; unit: Hypoglycemic Events
Units Other Than Participants: Hypoglycemic Events
Arm/Group | Nasal Glucagon
Number analyzed (Participants) | 14
Number analyzed (Hypoglycemic Events) | 33
Hypoglycemic Events
  Difficulty: opening the kit (Easy) | 6
  Difficulty: opening the kit (Very Easy) | 27
  Difficulty: instructions (Average) | 4
  Difficulty: instructions (Relatively Easy) | 1
  Difficulty: instructions (Easy) | 6
  Difficulty: instructions (Very Easy) | 22
  Difficulty: administering (Average) | 2
  Difficulty: administering (Easy) | 11
  Difficulty: administering (Very Easy) | 20
  Time to administer (<30 seconds) | 20
  Time to administer (30-<60 seconds) | 9
  Time to administer (1-<2 minutes) | 4
  Degree of satisfaction (Average) | 2
  Degree of satisfaction (Relatively Easy) | 1
  Degree of satisfaction (Easy) | 8
  Degree of satisfaction (Very Easy) | 22
  Compare to Injectable (Not Applicable) | 25
  Compare to Injectable (Much Easier) | 2
  Compare to Injectable (Easier) | 2
  Compare to Injectable (About the Same) | 4
  Ease to teach other (Easy) | 4
  Ease to teach other (Very Easy) | 29

3. Secondary Outcome: Percentage of Participants With Adverse Events Through the Nasal Score Questionnaire
Description: Adverse events solicited through the Nasal Score Questionnaire included: runny nose, nasal congestion (nostrils plugged), nasal itching, sneezing, watery eyes, itchy eyes, redness of eyes, itching of ears, itching of throat, and other.
  A summary of other non-serious AEs, and all SAE's, regardless of causality, is located in the Reported Adverse Events section.
Time Frame: Within 2 hours of full recovery from a hypoglycemic event
Population: Participants who received at least 1 dose of NG and experienced at least 1 hypoglycemic event.Participants from the GCP non-compliant site were considered ineligible and thus excluded from this population.
Measure: Number; unit: percentage of participants
Arm/Group | Nasal Glucagon
Number analyzed (Participants) | 14
percentage of participants | 100

4. Other Pre Specified Outcome: Change in Blood Glucose Level Over Time
Description: Glucometer-based measurements of blood glucose after the studied drug administration. The participants' change in blood glucose level from baseline (just prior to dosing or right after the study drug administration) was measured by the caregiver using a glucometer at 15, 30 and 45 minutes after NG administration. The change in glucose was calculated from each time point (15, 30 and 45 minutes) minus the baseline.
Time Frame: Baseline (just prior to dosing or right after study drug administration), 15, 30 and 45 minutes after drug administration for an episode of hypoglycemia
Population: Participants received at least 1 dose of the NG and experienced at least 1 hypoglycemic event. Participants from the GCP non-compliant site were considered ineligible and thus excluded from this population.
Measure: Mean (Standard Deviation); unit: milligram/deciliter (mg/dL)
Arm/Group | Nasal Glucagon
Number analyzed (Participants) | 14
milligram/deciliter (mg/dL)
  15 minutes drug administration | 58.2 (21.16)
  30 minutes drug administration | 106.8 (39.57)
  45 minutes drug administration | 124.1 (49.09)

ADVERSE EVENTS:
Description: All participants who received at least one dose of NG, including GCP non-compliance site.
  Adverse events were collected systematically using the Hypoglycemia Questionnaire.
Groups:
- Nasal Glucagon: 3 mg glucagon powder
Arm/Group | Nasal Glucagon
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 20/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nasal Glucagon (N=22)
Abdominal Pain Upper (Gastrointestinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Face Injury (Injury, poisoning and procedural complications) | 1 (4)
Fatigue (General disorders) | 1 (1)
Headache (General disorders) | 14 (26)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Incomplete Dose Administered (Investigations) | 1 (1)
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 19 (41) — Hypoglycemia Questionnaire vocabulary name.
Nausea (Gastrointestinal disorders) | 6 (10)
Paranasal Sinus Hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Product Taste Abnormal (General disorders) | 1 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Somnolence (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Watery Eyes (Eye disorders) | 18 (37) — Hypoglycemia Questionnaire vocabulary name.
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Participants from non-GCP compliant site were excluded from the analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less